CLINICAL TRIAL: NCT02683772
Title: The Evaluation of the Astral VAPS AutoEPAP Treatment Algorithm
Brief Title: Astral VAPS AutoEPAP Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MA-15-12-15
Record Dates: First submitted 2016-02-03; First posted 2016-02-17 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Upper Airway Obstruction; Respiratory Insufficiency; Respiratory Failure
Keywords: NIV, NIPPV, ventilation
MeSH Terms: conditions — Airway Obstruction; Respiratory Insufficiency; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients were masked to the mode of treatment. The Core Lab was masked to the mode of treatment for all patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- iVAPS with AutoEPAP (Experimental): This is a crossover study. During overnight PSG, Astral device will be set using iVAPS with AutoEPAP on the first night, and on iVAPS with manual EPAP on the second night.
  Interventions: Device: Astral
- iVAPS with manual EPAP (Active Comparator): This is a crossover study. During overnight PSG, Astral device will be set using iVAPS with manual EPAP on the first night, and on iVAPS with AutoEPAP on the second night.
  Interventions: Device: Astral

INTERVENTIONS:
Device: Astral — Astral ventilator

SUMMARY:
Patients with chronic respiratory failure such as those associated with Chronic Obstructive Pulmonary Disease (COPD), Obesity Hypoventilation Syndrome (OHS), Obstructive Sleep Apnea (OSA) or Neuromuscular Disease (NMD) are increasingly managed with domiciliary non-invasive positive pressure ventilation (NIPPV). The aim of this study is to now compare the Automatic Expiratory Positive Airway Pressure (AutoEPAP) algorithm with a fixed manual EPAP in iVAPS mode on an Astral mixed mode ventilator. It is proposed that the automatic settings of AutoEPAP will be as effective at managing respiratory failure and upper airway obstruction (UAO) as manual EPAP on the Astral device. Specifically demonstrating that the AutoEPAP function is as effective at treating UAO as manual EPAP.

ELIGIBILITY:
Inclusion criteria for the study are:

1. Participant has ability to provide written informed consent
2. Participants aged ≥18 years old
3. Participant has documented respiratory failure (e.g. sleep hypoventilation with historical PtCO2 increase ≥ 10mmHg) and/or daytime hypercapnia (>45 mmHg)
4. Participant is currently using non-invasive positive pressure ventilation in ST or VAPS mode for ≥ 3 months
5. Participants with a previously documented AHI ≥ 5/hr
6. Participants with a recently (≤ 12 months ago) reviewed EPAP setting

Exclusion criteria for the study are:

1. Participants are not compliant on NIPPV (e.g. < 4 hr/night)
2. Participants who are pregnant
3. Participants on oxygen therapy ≥5 L/min
4. Participants with an invasive interface (e.g. tracheostomy)
5. Participants who have had an acute exacerbation within the last 3 months that resulted in a hospitalisation
6. Participants who are acutely ill, medically complicated or who are medically unstable
7. Participants in whom NIPPV therapy is otherwise medically contraindicated
8. Participants who have had surgery of the upper airway, nose, sinus, or middle ear within the previous 90 days
9. Participants with untreated, non-OSA sleep disorders, including but not limited to; insomnia, periodic limb movement syndrome, or restless legs syndrome.
10. Participants who have the following pre-existing conditions: severe bullous lung disease, recurrent pneumothorax or pneumomediastinum, cerebrospinal fluid leak, recent cranial surgery or trauma.
11. Participant does not comprehend English
12. Participant is unable or unwilling to provide written informed consent
13. Participant is physically and/or mentally unable to comply with the protocol
14. Participant is not suitable to participate in the trial for any other reason in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Wolfe, MD, Principal Investigator — Northwestern Medical Center
Locations (5):
- United States (5):
  - University of California, San Diego, La Jolla, California
  - National Jewish Health, Denver, Colorado
  - Lisa F. Wolfe, MD, Chicago, Illinois
  - Temple University, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Budweiser S, Jorres RA, Riedl T, Heinemann F, Hitzl AP, Windisch W, Pfeifer M. Predictors of survival in COPD patients with chronic hypercapnic respiratory failure receiving noninvasive home ventilation. Chest. 2007 Jun;131(6):1650-8. doi: 10.1378/chest.06-2124. PMID 17565016
- [Background] Masa JF, Celli BR, Riesco JA, Hernandez M, Sanchez De Cos J, Disdier C. The obesity hypoventilation syndrome can be treated with noninvasive mechanical ventilation. Chest. 2001 Apr;119(4):1102-7. doi: 10.1378/chest.119.4.1102. PMID 11296176
- [Background] Remmers JE, deGroot WJ, Sauerland EK, Anch AM. Pathogenesis of upper airway occlusion during sleep. J Appl Physiol Respir Environ Exerc Physiol. 1978 Jun;44(6):931-8. doi: 10.1152/jappl.1978.44.6.931. No abstract available. PMID 670014
- [Background] Ward S, Chatwin M, Heather S, Simonds AK. Randomised controlled trial of non-invasive ventilation (NIV) for nocturnal hypoventilation in neuromuscular and chest wall disease patients with daytime normocapnia. Thorax. 2005 Dec;60(12):1019-24. doi: 10.1136/thx.2004.037424. PMID 16299118
- [Background] Laghi F, Tobin MJ. Disorders of the respiratory muscles. Am J Respir Crit Care Med. 2003 Jul 1;168(1):10-48. doi: 10.1164/rccm.2206020. PMID 12826594
- [Derived] Suh ES, Murphy PB. Auto-titration of EPAP during NIV: A better night's sleep? Respirology. 2019 Dec;24(12):1132-1133. doi: 10.1111/resp.13587. Epub 2019 May 23. No abstract available. PMID 31120585
- [Derived] Orr JE, Coleman J, Criner GJ, Sundar KM, Tsai SC, Benjafield AV, Crocker ME, Willes L, Malhotra A, Owens RL, Wolfe LF. Automatic EPAP intelligent volume-assured pressure support is effective in patients with chronic respiratory failure: A randomized trial. Respirology. 2019 Dec;24(12):1204-1211. doi: 10.1111/resp.13546. Epub 2019 Apr 22. PMID 31012225

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 43 patients consented for this study. One patient did not meet criteria. 42 patients were randomized and began the first study PSG night. 3 patients were found to be ineligible due to I/E criteria not met. Site erroneously placed patient on ST mode for one of the PSG study nights. Thus, there were 38 patients that were analyzed.
Groups:
- iVAPS With AutoEPAP, Then iVAPS With Manual EPAP: This is a crossover study. After randomization, patients in this arm will receive overnight PSG iVAPS with AutoEPAP first, and the second night iVAPS with manual EPAP. Therapy will be delivered using the clinical trial device, Astral. At least 4 hours of recording will be required.
- iVAPS With Manual EPAP, Then iVAPS With AutoEPAP: This is a crossover study. After randomization, patients in this arm will receive overnight PSG iVAPS with manual EPAP first, and the second night iVAPS with AutoEPAP. Therapy will be delivered using the clinical trial device, Astral. At least 4 hours of recording will be required.
Period: Overall Study
Arm/Group | iVAPS With AutoEPAP, Then iVAPS With Manual EPAP | iVAPS With Manual EPAP, Then iVAPS With AutoEPAP
Started | 15 | 23
Completed | 15 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This is a crossover study. There were 42 patients enrolled in total. 38 patients met the definition of evaluable. These 38 participated in both 'Group A' and 'Group B' intervention assignments. All Baseline characteristics are summarized for these 38 evaluable patients.
Groups:
- Study Total: This is a crossover study. There were 42 patients enrolled in total. 38 patients met the definition of evaluable. These 38 participated in both 'Group A' and 'Group B' intervention assignments. All Baseline characteristics are summarized for these 38 evaluable patients.
Arm/Group | Study Total
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.33 (16.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 8
  White | 23
  More than one race | 0
  Unknown or Not Reported | 5
BMI [Mean (Standard Deviation); unit: kg/m^2] | 34.41 (9.84)

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Desaturation Index 4% (ODI4%)
Description: Mean paired difference AutoEPAP-manual EPAP: Comparison of Oxygen Desaturation Index 4% (ODI4%) values between groups by using mean ODI4% (#events/hour). A cross-over analysis was generated to investigate the influence of a possible period effect on the primary endpoint, paired change in ODI4% between Auto and manual EPAP
Time Frame: Overnight, up to 8 hrs on nights 1 and 2
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: events per hour
Groups:
- iVAPS With AutoEPAP: This is a crossover study. There were 42 patients enrolled in total. 38 patients met the definition of evaluable. These 38 participated in both iVAPS with AutoEPAP and iVAPS with manual EPAP intervention assignments. All Baseline characteristics are summarized for these 38 evaluable patients.
- iVAPS With Manual EPAP: This is a crossover study. There were 42 patients enrolled in total. 38 patients met the definition of evaluable. These 38 participated in both iVAPS wtih AutoEPAP and iVAPS with manual EPAP intervention assignments. All Baseline characteristics are summarized for these 38 evaluable patients.
Arm/Group | iVAPS With AutoEPAP | iVAPS With Manual EPAP
Number analyzed (Participants) | 38 | 38
events per hour | 3.16 (5.67) | 7.61 (18.87)
Statistical Analysis 1: Comparison: iVAPS With AutoEPAP vs iVAPS With Manual EPAP; Test type: Non-Inferiority — The method proposed for this analysis was a one-sided paired t-test using a significance level of 0.05 and a non-inferiority margin of 2 events/hour; p = 0.0134, t-test, 1 sided; Mean Difference (Final Values) = -4.45, Standard Deviation 17.23

2. Secondary Outcome: Sleep Efficiency (%)
Description: To assess sleep efficacy between groups by using rapid eye movement sleep (REM) (% of total sleep time)
Time Frame: Overnight, up to 8 hrs on nights 1 and 2
Measure: Mean (Standard Deviation); unit: percentage of total sleep time
Groups:
- iVAPS With AutoEPAP: Astral device will be set using iVAPS with autoEPAP for the overnight PSG
  Astral: Astral ventilator
- iVAPS With Manual EPAP: Astral device will be set using iVAPS with manual EPAP during overnight PSG
  Astral: Astral ventilator
Arm/Group | iVAPS With AutoEPAP | iVAPS With Manual EPAP
Number analyzed (Participants) | 38 | 38
percentage of total sleep time | 73.70 (16.41) | 73.89 (19.05)

3. Secondary Outcome: Apnea Hypopnea Index (AHI)
Description: To assess sleep-breathing parameters between groups using mean AHI (#events/hour)
Time Frame: Overnight, up 8 hrs on night 1 and 2
Population: Analysis population in each arm/group is based on the total number of participants receiving each intervention over two separate nights.
Measure: Mean (Standard Deviation); unit: events per hour
Groups:
- iVAPS With AutoEPAP: This is a crossover study. After randomization, patients in this arm will receive overnight PSG iVAPS with AutoEPAP first, and the second night iVAPS with manual EPAP. Therapy will be delivered using the clinical trial device, Astral. At least 4 hours of recording will be required.
- iVAPS With Manual EPAP: This is a crossover study. After randomization, patients in this arm will receive overnight PSG iVAPS with manual EPAP first, and the second night iVAPS with AutoEPAP. Therapy will be delivered using the clinical trial device, Astral. At least 4 hours of recording will be required.
Arm/Group | iVAPS With AutoEPAP | iVAPS With Manual EPAP
Number analyzed (Participants) | 38 | 38
events per hour | 4.71 (5.55) | 7.84 (15.39)

4. Secondary Outcome: Nadir Arterial Oxygen Saturation (SpO2)
Description: To assess Sleep-breathing parameters between groups using mean SpO2 (%)
Time Frame: Overnight, up 8 hrs on night 1 and 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | iVAPS With AutoEPAP | iVAPS With Manual EPAP
Number analyzed (Participants) | 38 | 38
percentage of oxygen saturation | 94.24 (2.36) | 94.53 (2.78)

5. Secondary Outcome: Arterial Carbon Dioxide (PCO2)
Description: To assess Sleep-breathing parameters between groups using mean PCO2 (mmHg)
Time Frame: Overnight, up 8 hrs on night 1 and 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milimeters of mercury
Arm/Group | iVAPS With AutoEPAP | iVAPS With Manual EPAP
Number analyzed (Participants) | 38 | 38
milimeters of mercury | 45.49 (6.62) | 45.38 (7.17)

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected for each patient enrolled into the study. AE data was collected from signing of Informed Consent Form until the patient's final completion date (PSG #2).
Groups:
- iVAPS With AutoEPAP; iVAPS With Manual EPAP: This is a crossover study. There were 42 patients randomized in total. 38 patients met the definition of evaluable. These 38 participated in both iVAPS with AutoEPAP and iVAPS with manual EPAP intervention assignments. Adverse Event data were collected for all 42 enrolled patients.
Arm/Group | iVAPS With AutoEPAP | iVAPS With Manual EPAP
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 1/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iVAPS With AutoEPAP (N=42) | iVAPS With Manual EPAP (N=42)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Patient woke up with an asthma exacerbation at 4:37am. Patient utilized her normal home routine treatment. This event was determined to be 'not related' to the device or study treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-06-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT02683772/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-23): https://cdn.clinicaltrials.gov/large-docs/72/NCT02683772/SAP_001.pdf